CLINICAL TRIAL: NCT06517732
Title: Prospective, Observational, Multicenter Study to Collect in a Real-world populatIon Data on the Treatment Pattern of Secukinumab in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (HS) in Routine Clinical Practice in the Russian Federation (ANIMA-R)
Brief Title: Study to Collect in a Real-world populatIon Data on the Treatment Pattern of Secukinumab in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (HS) in Routine Clinical Practice in the Russian Federation
Acronym: ANIMA-R
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MRU01
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; HS; real-world data; secukinumab
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Secukinumab: Patients prescribed with secukinumab in the treatment of Hidradenitis Suppurativa
  Interventions: Other: Secukinumab

INTERVENTIONS:
Other: Secukinumab — This is an observational study. There is no treatment allocation. The decision to initiate secukinumab will be based solely on clinical judgement.

SUMMARY:
ANIMA-R is an observational, prospective, non-interventional, multicenter study to assess real-world effectiveness of secukinumab in the treatment of Hidradenitis Suppurativa (HS).

DETAILED DESCRIPTION:
The index date will be the date of secukinumab initiation. During the study, data will be collected from patients receiving routine secukinumab treatment, which is representative of the actual patient population.

The attending physician will decide whether to prescribe secukinumab based on the approved instructions for medical use in a routine clinical setting, regardless of the patient's participation in a non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provide written informed consent form (ICF) to participate in the study.
2. Male and female.
3. ≥ 18 years old.
4. Diagnosis of moderate or severe HS (Hurley stage and IHS4).
5. Patient who initiated treatment with secukinumab no longer than 4 weeks prior to written ICF.
6. Decision for secukinumab prescription was made by the attending physician according to the approved national label during routine clinical practice, regardless of study participation.

Exclusion Criteria:

1. Any medical or psychological condition that may prevent the study participation, based on practitioners' decision-making.
2. Participation in an ongoing clinical trial.
3. Known or suspected severe hypersensitivity for secukinumab, formulation excipients, or injection device components (i.e., latex).
4. Clinically significant infection exacerbation, including active tuberculosis.
5. Patients with active inflammatory bowel disease (IBD).
6. Age <18 years.
7. Pregnancy and breastfeeding.
8. Patients who received any vaccine within 4 weeks prior to secukinumab initiation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe Hidradenitis Suppurativa commencing treatment with secukinumab
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving 55% reduction in IHS4 (IHS4-55) | 12 months
  The International Hidradenitis Suppurativa Severity Scoring System (IHS4) allows for a dynamic assessment of the disease severity both in clinical studies and in real-world clinical setting. The IHS4 is determined by counting nodules, abscesses, and draining tunnels (fistulae/sinuses). IHS4 (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or lower indicates a mild stage of hidradenitis suppurativa, a score of 4-10 indicates a moderate stage, and a score of 11 or higher indicates a severe stage of the disease. The IHS4 severity scoring system assumes that the presence of a draining tunnel (fistula/sinus) is sufficient to classify a case as at least moderate.

SECONDARY OUTCOMES:
Proportion of patients receiving HS-specific concomitant treatments in combination with secukinumab | 12 months
  Proportion of patients receiving Hidradenitis Suppurativa (HS)-specific concomitant treatments in combination with secukinumab
Time of initiation of concomitant medication | 12 months
  Time of initiation of concomitant medication (before or after the initiation of secukinumab).
Duration of treatment with concomitant medication | 12 months
  Duration of treatment with concomitant medication of secukinumab
Number, type, and outcome of surgical interventions | 12 months
  Number, type, and outcome of surgical interventions (minor and major surgical excision; inpatient, outpatient, or self-treatment at home)
Timepoint of and reason for surgical intervention | 12 months
  Timepoint of and reason for surgical intervention.
Duration of discontinuation/pause of secukinumab treatment before surgery | 12 months
  Duration of discontinuation/pause of secukinumab treatment before surgery
Duration of discontinuation/pause of secukinumab treatment after surgery | 12 months
  Duration of discontinuation/pause of secukinumab treatment after surgery
Surgery outcome | 12 months
  Surgery outcome by type of wound healing, pain relief and discontinuation or continuation of secukinumab.
Outcome of surgery and adverse events stratified by secukinumab management | 12 months
  Outcome of surgery (healing, pain relief) and adverse events (i.e., infections) stratified by secukinumab management (continuation or discontinuation).
Predictors of treatment response | 12 months
  Listing of predictors of treatment response
Proportion of patients achieving 75% reduction in IHS4 (IHS4-75) and 100% reduction in IHS4 (IHS4-100) | Month 6, month 12
  The International Hidradenitis Suppurativa Severity Scoring System (IHS4) allows for a dynamic assessment of the disease severity both in clinical studies and in real-world clinical setting. The IHS4 is determined by counting nodules, abscesses, and draining tunnels (fistulae/sinuses). IHS4 (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4]. A score of 3 or lower indicates a mild stage of hidradenitis suppurativa, a score of 4-10 indicates a moderate stage, and a score of 11 or higher indicates a severe stage of the disease. The IHS4 severity scoring system assumes that the presence of a draining tunnel (fistula/sinus) is sufficient to classify a case as at least moderate.
Lesion spread | Baseline, month 6, month 12
  Lesion spread (defined as total abscess and inflammatory nodule count (AN) or draining fistula in a body region not seen at baseline) assessed by number, type, and localization of HS lesions
Mean change of nodule count | Month 6, month 12
  Mean reduction of nodule count

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Russia (15):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kaliningrad
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yakutsk

IPD SHARING:
Plan to Share IPD: No